CLINICAL TRIAL: NCT03956992
Title: Effects of a Hydroxyapatite-based Mouth Gel on Calcium Content of Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Joachim Enax (Industry)
Responsible Party: Sponsor-Investigator, Dr. Joachim Enax, Senior Scientist Oral Care, Dr. Kurt Wolff GmbH & Co. KG
Organization: Dr. Kurt Wolff GmbH & Co. KG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dr. Kurt Wolff
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mouth gel (Experimental): A mouth gel with hydroxyapatite
  Interventions: Other: Mouth gel

INTERVENTIONS:
Other: Mouth gel — Stop using the mouth gel

SUMMARY:
The aim of this pilot study is to analyze if a hydroxyapatite-containing mouth gel has an influence on the calcium content of plaque.

DETAILED DESCRIPTION:
>= 20 subjects (7-11 years) use the hydroxyapatite-containing mouth gel for 3 days (3x per day); without using any other oral care product at this time. A dentist applies the gel on all teeth. At baseline and after 3 days plaque will be collected from buccal and labial surfaces (except surfaces with tartar). A "split-mouth" concept will be used:

Subjects in group A:

Baseline plaque collection: quadrant 1 and 4 Plaque collection after 3 days: quadrant 2 and 3

Subjects in group B:

Baseline plaque collection: quadrant 2 and 3 Plaque collection after 3 days: quadrant 1 and 4 (The time between last application of the gel and plaque collection will be 1 h) The plaque will be dried and afterwards the calcium content of the plaque will be quantitively analyzed by atomic absorption spectroscopy (AAS).

For all subjects: Calcium contents of plaque at baseline and after 3 days application will be compared by statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys (7-11 years)
* Visible plaque
* >= 4 teeth
* Good overall health

Exclusion Criteria:

* Allergic to one or more ingredients of the mouth gel
* Medication intake (e.g. antibiotics)
* Any other reason that, in the opinion of the investigator, disqualifies the subject from participating in the study

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Calcium content of plaque | 3 days
  Analysis by atomic absorption spectroscopy (AAS)

CONTACTS AND LOCATIONS:
Overall Officials: Henny Sudradjat, Principal Investigator — Department for Dentistry, Health Care Center, Braunschweig, Germany
Locations (1):
- Health department, Bali, Kebon Padangan, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw L, Murray JJ, Burchell CK, Best JS. Calcium and phosphorus content of plaque and saliva in relation to dental caries. Caries Res. 1983;17(6):543-8. doi: 10.1159/000260715. No abstract available. PMID 6580080